CLINICAL TRIAL: NCT04599855
Title: A Randomized, Double-blind, Multicenter, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Esketamine Nasal Spray, Administered as Monotherapy, in Adult Participants With Treatment-resistant Depression
Brief Title: A Study of Esketamine Nasal Spray, Administered as Monotherapy, in Adult Participants With Treatment-resistant Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108741; 54135419TRD4005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-10-21; First posted 2020-10-23 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Treatment-Resistant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Esketamine 56 Milligram (mg) (Experimental): Participants will receive nasal spray treatment with esketamine 56 mg twice a week for 4 weeks. Participants may participate in an open-label treatment/observation phase, following completion of the double-blind treatment phase assessments (which includes the Day 28 Montgomery-Asberg Depression Rating Scale [MADRS] assessment).
  Interventions: Drug: Esketamine 56 mg
- Esketamine 84 mg (Experimental): Participants will receive nasal spray treatment with esketamine 84 mg twice a week for 4 weeks. Participants may participate in an open-label treatment/observation phase, following completion of the double-blind treatment phase assessments (which includes the Day 28 MADRS assessment).
  Interventions: Drug: Esketamine 84 mg
- Placebo (Experimental): Participants will receive nasal spray treatment with placebo twice a week for 4 weeks. Participants may participate in an open-label treatment/observation phase, following completion of the double-blind treatment phase assessments (which includes the Day 28 MADRS assessment).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esketamine 56 mg — Esketamine 56 mg will be self administered as nasal spray.
  Other Names: JNJ-54135419
  Arms: Esketamine 56 Milligram (mg)
Drug: Esketamine 84 mg — Esketamine 84 mg will be self administered as nasal spray.
  Other Names: JNJ-54135419
  Arms: Esketamine 84 mg
Drug: Placebo — Matching placebo will be self administered as nasal spray.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of each individual dose of esketamine nasal spray, 56 milligram (mg) and 84 mg, compared with placebo nasal spray in improving depressive symptoms in participants with treatment resistant depression (TRD), as assessed by the change from baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) total score from Day 1 (prerandomization) to the end of the 4 week double-blind treatment phase (Day 28).

ELIGIBILITY:
Inclusion Criteria:

* Participant must meet the Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5) diagnostic criteria for single-episode MDD or recurrent MDD, without psychotic features, based upon clinical assessment and confirmed by the MINI. Participants 65 years of age or older must have had the first onset of depression prior to 55 years of age
* Participant must have had nonresponse (<=25% improvement) to >=2 oral antidepressant treatments in the current episode of depression, assessed using the MGH-ATRQ, and confirmed by documented records (example, medical/pharmacy/prescription records or a letter from a treating physician)
* Participant must have an Inventory of Depressive Symptomatology-Clinician rated, 30-item (IDS-C30) total score of >=34
* The participant's current major depressive episode, depression symptom severity, and antidepressant treatment response in the current depressive episode, must be confirmed by the State vs. Trait, Assessibility, Face Validity, Ecological Validity, Rule of Three P's (SAFER) Interview
* Participant must be medically stable on the basis of physical examination, medical history, vital signs (including blood pressure), and 12-lead electrocardiogram (ECG) performed in the screening phase. If there are any abnormalities that are not specified in the inclusion and exclusion criteria, the determination of their clinical significance must be determined by the investigator and recorded in the participant's source documents and initiated by the investigator
* Participant must be medically stable on the basis of clinical laboratory tests performed in the screening phase. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator: (a) Participants with a pre-existing history of thyroid disease/disorder who are treated with thyroid hormones must be on a stable dosage for 3 months prior to the start of the screening phase; (b) For any participant (regardless of thyroid history), if the thyroid-stimulating hormone (TSH) value is out of range, a free thyroxine (FT4) will be conducted. If the FT4 value is abnormal and considered to be clinically significant (after discussion with the medical monitor), the participant is not eligible
* Participant must be comfortable with self-administration of nasal spray medication and be able to follow the nasal spray administration instructions provided

Exclusion Criteria:

* The participant has used ketamine/esketamine (lifetime)
* The participant's depressive symptoms have previously demonstrated nonresponse to an adequate course of treatment with electroconvulsive therapy (ECT) in the current major depressive episode, defined as at least 7 treatments with unilateral/bilateral ECT
* Participant has received vagal nerve stimulation (VNS) or has received deep brain stimulation (DBS) in the current episode of depression
* Participant has a current or history of seizures (uncomplicated childhood febrile seizures with no sequelae are not exclusionary)
* Participant has any anatomical or medical condition that, per the investigator's clinical judgment based on assessment, may impede delivery or absorption of nasal spray study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (54):
- United States (54):
  - UAB Department of Psychiatry and Behavioral Neurobiology, Birmingham, Alabama
  - UAB Huntsville Regional Medical Campus, Huntsville, Alabama
  - Preferred Research Partners, Little Rock, Arkansas
  - Behavioral Research Specialists LLC, Glendale, California
  - CalNeuro Research, Los Angeles, California
  - Pacific Research Partners, Oakland, California
  - Anderson Clinical Research, Redlands, California
  - University of California at San Diego, San Diego, California
  - Artemis Institute for Clinical Research, San Diego, California
  - UCSF Nancy Friend Pritzker Psychiatry Building, San Francisco, California
  - Velocity Clinical Research, Santa Ana, California
  - CMB Clinical Trials, Santee, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Accel Research Sites, Lakeland, Florida
  - APG Research LLC, Orlando, Florida
  - USF, Department of Psychiatry and Behavioral Neurosciences, Tampa, Florida
  - Neuroscience Research Institute, West Palm Beach, Florida
  - Atlanta Behavioral Research, LLC, Atlanta, Georgia
  - Psych Atlanta, P.C., Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Chicago Research Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Joliet Center for Clinical Research, Joliet, Illinois
  - Pillar Clinical Research, LLC, Lincolnwood, Illinois
  - Psychiatric Medicine Associates LLC, Skokie, Illinois
  - Ascension via Christi Research, Wichita, Kansas
  - University of Kansas School of Medicine, Wichita, Kansas
  - Sheppard Pratt Health System, Baltimore, Maryland
  - CBH Health, Gaithersburg, Maryland
  - Copley Clinical, Boston, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Rochester Center for Behavioral Medicine (RCBM), Rochester Hills, Michigan
  - Midwest Research Group - St. Charles Psychiatric Associates, Saint Charles, Missouri
  - Clinilabs, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Ohio State University, Columbus, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Paradigm Research Professionals, LLC, Oklahoma City, Oklahoma
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - The Warren Alpert Medical School of Brown University - Butler Hospital, Providence, Rhode Island
  - BioBehavioral Research of Austin PC, Austin, Texas
  - Relaro Medical Trials, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Brain Health Consultants and TMS Center, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - University of Virginia Center for Psychiatric Clinical Research, Charlottesville, Virginia

REFERENCES:
- [Derived] Janik A, Qiu X, Lane R, Popova V, Drevets WC, Canuso CM, Macaluso M, Mattingly GW, Shelton RC, Zajecka JM, Fu DJ. Esketamine Monotherapy in Adults With Treatment-Resistant Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2025 Sep 1;82(9):877-887. doi: 10.1001/jamapsychiatry.2025.1317. PMID 40601310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with recurrent or single (duration greater than or equal to [>=] 2 years) episode major depressive disorder (DSM-5 criteria) without psychotic features who experienced inadequate response (less than or equal to [<=] 25 percent [%] improvement) to >=2 oral antidepressants during the current depressive episode were randomized in the study.
Groups:
- Placebo: In the double-blind (DB) phase, participants received placebo nasal spray (matching to esketamine) twice a week for 4 weeks on Days 1, 4, 8, 11, 15, 18, 22, and 25. After completion of the DB phase (including Day 28 visit), participants opted to enter the open-label (OL) phase (treatment/observation phase). Participants who opted OL treatment phase received esketamine 56 milligrams (mg) nasal spray on Day 28 regardless of the treatment assignment in the DB phase and received subsequent doses at the same or adjusted (56 mg or 84 mg) dose level based on efficacy and tolerability with dosing frequency: twice weekly from Weeks 5 to 8 followed by once weekly from Weeks 9 to 12 and then weekly or every other week from Weeks 13 to 16 based on clinical judgment and was individualized to the least frequent dosing to maintain remission/response. During this period participants were given the option to receive standard-of-care treatment for depression. Participants who opted OL observation phase were only observed without esketamine nasal spray treatment but received standard-of-care treatment for depression. All participants underwent 1-week follow-up phase for safety assessment after their last dose of study treatment in DB or OL treatment phase.
- Esketamine 56 mg: In the DB phase, participants received esketamine 56 mg nasal spray twice a week for 4 weeks on Days 1, 4, 8, 11, 15, 18, 22, and 25. After completion of the DB phase (including Day 28 visit), participants opted to enter the OL phase (treatment/observation phase). Participants who opted OL treatment phase received esketamine 56 mg nasal spray on Day 28 regardless of the treatment assignment in the DB phase and received subsequent doses at the same or adjusted (56 mg or 84 mg) dose level based on efficacy and tolerability with dosing frequency: twice weekly from Weeks 5 to 8 followed by once weekly from Weeks 9 to 12 and then weekly or every other week from Weeks 13 to 16 based on clinical judgment and was individualized to the least frequent dosing to maintain remission/response. During this period participants were given the option to receive standard-of-care treatment for depression. Participants who opted OL observation phase were only observed without esketamine nasal spray treatment but received standard-of-care treatment for depression. All participants underwent 1-week follow-up phase for safety assessment after their last dose of study treatment in DB or OL treatment phase.
- Esketamine 84 mg: In the DB phase, participants received esketamine 84 mg nasal spray twice a week for 4 weeks on Days 1, 4, 8, 11, 15, 18, 22, and 25. After completion of the DB phase (including Day 28 visit), participants opted to enter the OL phase (treatment/observation phase). Participants who opted OL treatment phase received esketamine 56 mg nasal spray on Day 28 regardless of the treatment assignment in the DB phase and received subsequent doses at the same or adjusted (56 mg or 84 mg) dose level based on efficacy and tolerability with dosing frequency: twice weekly from Weeks 5 to 8 followed by once weekly from Weeks 9 to 12 and then weekly or every other week from Weeks 13 to 16 based on clinical judgment and was individualized to the least frequent dosing to maintain remission/response. During this period participants were given the option to receive standard-of-care treatment for depression. Participants who opted OL observation phase were only observed without esketamine nasal spray treatment but received standard-of-care treatment for depression. All participants underwent 1-week follow-up phase for safety assessment after their last dose of study treatment in DB or OL treatment phase.
Period: Double Blind Period (Day 1 to Day 28)
Arm/Group | Placebo | Esketamine 56 mg | Esketamine 84 mg
Started | 250 | 106 | 121
Treated | 250 | 105 | 121
Completed | 238 | 101 | 107
Not Completed | 12 | 5 | 14
Not completed — Withdrawal by Subject | 5 | 2 | 5
Not completed — Adverse Event | 2 | 1 | 5
Not completed — Lack of Efficacy | 2 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Other | 1 | 0 | 1
Not completed — Randomized but not treated | 0 | 1 | 0
Period: Period Title: OL Period (Week 5 to 16)
Arm/Group | Placebo | Esketamine 56 mg | Esketamine 84 mg
Started | 237 | 99 | 106
Participants Who Entered OL Treatment Phase | 237 | 99 | 105
Participants Who Entered OL Observation Phase | 0 | 0 | 1
Completed | 204 | 87 | 95 (Included one participant who entered OL observation phase.)
Not Completed | 33 | 12 | 11
Not completed — Withdrawal by Subject | 8 | 5 | 6
Not completed — Lack of Efficacy | 10 | 3 | 2
Not completed — Adverse Event | 4 | 2 | 1
Not completed — Lost to Follow-up | 4 | 1 | 2
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Other | 5 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants (participants who met and did not meet nonresponse criteria) who received at least 1 dose of DB study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Esketamine 56 mg | Esketamine 84 mg | Total
Number analyzed (Participants) | 250 | 105 | 121 | 476
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 229 | 95 | 107 | 431
  >=65 years | 21 | 10 | 14 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.4 (13.72) | 45.1 (13.92) | 45.1 (14.75) | 45.3 (14.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 60 | 77 | 284
  Male | 103 | 45 | 44 | 192
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 9 | 8 | 42
  Not Hispanic or Latino | 221 | 95 | 112 | 428
  Unknown or Not Reported | 4 | 1 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 6 | 3 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 17 | 7 | 11 | 35
  White | 217 | 91 | 102 | 410
  More than one race | 6 | 1 | 2 | 9
  Unknown or Not Reported | 4 | 1 | 0 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 250 | 105 | 121 | 476

OUTCOME MEASURES:

1. Primary Outcome: Double-blind Treatment Phase: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score From Day 1 (Pre-randomization) to Day 28
Description: The MADRS was a clinician-rated scale designed to measure depression severity and detect changes due to antidepressant treatment. The scale consisted of 10 items, each of which was scored from 0 (item not present or normal) to 6 (severe or continuous presence of symptoms). MADRS total score was the sum of scores from individual question items, which ranged from 0 to 60, higher scores represented a more severe condition. The MADRS evaluated apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, inability to feel (interest level), pessimistic thoughts, and suicidal thoughts. Negative change in MADRS total score indicated improvement.
Time Frame: Day 1 (pre-randomization) to Day 28 (end of DB treatment phase)
Population: Full efficacy analysis set included all randomized participants who met nonresponse criteria and received at least 1 dose of DB study intervention. Here 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- DB: Placebo: In the double-blind (DB) phase, participants received placebo nasal spray (matching to esketamine) twice a week for 4 weeks on Days 1, 4, 8, 11, 15, 18, 22, and 25. All participants underwent 1-week follow-up phase for safety assessment after their last dose of study treatment in DB phase.
- DB: Esketamine 56 mg: In the DB phase, participants received esketamine 56 mg nasal spray twice a week for 4 weeks on Days 1, 4, 8, 11, 15, 18, 22, and 25. All participants underwent 1-week follow-up phase for safety assessment after their last dose of study treatment in DB phase.
- DB: Esketamine 84 mg: In the DB phase, participants received esketamine 84 mg nasal spray twice a week for 4 weeks on Days 1, 4, 8, 11, 15, 18, 22, and 25. All participants underwent 1-week follow-up phase for safety assessment after their last dose of study treatment in DB phase.
Arm/Group | DB: Placebo | DB: Esketamine 56 mg | DB: Esketamine 84 mg
Number analyzed (Participants) | 185 | 82 | 89
Score on a scale | -7.0 (10.07) | -12.7 (11.82) | -13.9 (11.89)
Statistical Analysis 1: Comparison: DB: Placebo vs DB: Esketamine 56 mg; Test type: Superiority; p < 0.001, Mixed model for repeated measures; least square (LS) means difference = -5.1, 95% CI 2-sided [-7.91 to -2.33], Standard Error of Mean 1.42
Statistical Analysis 2: Comparison: DB: Placebo vs DB: Esketamine 84 mg; Test type: Superiority; p < 0.001, Mixed model for repeated measures; LS means difference = -6.8, 95% CI 2-sided [-9.48 to -4.07], Standard Error of Mean 1.38

2. Secondary Outcome: Double-blind Treatment Phase: Change in MADRS Total Score From Day 1 (Pre-randomization) to Day 2 (24 Hours Post First Dose on Day 1)
Description: as for outcome 1
Time Frame: Day 1 (pre-randomization) to Day 2 of DB treatment phase (24 hours post first dose on Day 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | DB: Placebo | DB: Esketamine 56 mg | DB: Esketamine 84 mg
Number analyzed (Participants) | 195 | 84 | 93
Score on a scale | -9.7 (10.27) | -13.9 (10.15) | -13.0 (9.68)
Statistical Analysis 1: Comparison: DB: Placebo vs DB: Esketamine 56 mg; Test type: Superiority; p = 0.004, Mixed model for repeated measures; LS means difference = -3.8, 95% CI 2-sided [-6.29 to -1.22], Standard Error of Mean 1.29
Statistical Analysis 2: Comparison: DB: Placebo vs DB: Esketamine 84 mg; Test type: Superiority; p = 0.006, Mixed model for repeated measures; LS means difference = -3.4, 95% CI 2-sided [-5.89 to -1.00], Standard Error of Mean 1.24

ADVERSE EVENTS:
Time Frame: Double-blind (DB) phase: From Day 1 (post-dose) to Day 28; Open-label (OL) phase: From Week 5 to Week 16; Follow-up (FU) phase: Up to 1 week after last dose of study drug in DB phase (Week 5) or OL treatment phase (Week 17)
Description: All cause mortality:Randomized analysis set:all randomized participants; serious adverse events (AE)/other AE:DB:Safety analysis set(SAS):all randomized participants who received at least 1 dose of DB intervention; OL arms:OL analysis set:all participants who received at least 1 dose of OL esketamine; OL observation arm:Observation analysis set:all participants who entered observation phase but did not receive OL esketamine; FU:SAS. FU:All Participants arm: combined data of DB and OL per plan.
Groups:
- DB: Placebo: In the double-blind (DB) phase, participants received placebo nasal spray (matching to esketamine) twice a week for 4 weeks on Days 1, 4, 8, 11, 15, 18, 22, and 25.
- DB: Esketamine 56 mg: In the DB phase, participants received esketamine 56 mg nasal spray twice a week for 4 weeks on Days 1, 4, 8, 11, 15, 18, 22, and 25.
- DB: Esketamine 84 mg: In the DB phase, participants received esketamine 84 mg nasal spray twice a week for 4 weeks on Days 1, 4, 8, 11, 15, 18, 22, and 25.
- OL Treatment: Placebo to Esketamine: Participants who received placebo in DB phase were given a choice either to receive esketamine nasal spray treatment or were observed only without nasal spray treatment. Participants who opted OL treatment phase received esketamine 56 mg nasal spray on Day 28 regardless of the treatment assignment in the DB phase and received subsequent doses at the same or adjusted (56 mg or 84 mg) dose level based on efficacy and tolerability with dosing frequency: twice weekly from Weeks 5 to 8 followed by once weekly from Weeks 9 to 12 and then weekly or every other week from Weeks 13 to 16 based on clinical judgment and was individualized to the least frequent dosing to maintain remission/response. During this period participants were given the option to receive standard-of-care treatment for depression. As planned, OL phase adverse events analysis was performed by treatment groups assigned in the DB phase, irrespective of the OL phase adjusted doses.
- OL Treatment: Esketamine 56 mg to Esketamine: Participants who received esketamine 56 mg in DB phase were given a choice either to receive esketamine nasal spray treatment or were observed only without nasal spray treatment. Participants who opted OL treatment phase received esketamine 56 mg nasal spray on Day 28 regardless of the treatment assignment in the DB phase and received subsequent doses at the same or adjusted (56 mg or 84 mg) dose level based on efficacy and tolerability with dosing frequency: twice weekly from Weeks 5 to 8 followed by once weekly from Weeks 9 to 12 and then weekly or every other week from Weeks 13 to 16 based on clinical judgment and was individualized to the least frequent dosing to maintain remission/response. During this period participants were given the option to receive standard-of-care treatment for depression. As planned, OL phase adverse events analysis was performed by treatment groups assigned in the DB phase, irrespective of the OL phase adjusted doses.
- OL Treatment: Esketamine 84 mg to Esketamine: Participants who received esketamine 84 mg in DB phase were given a choice either to receive esketamine nasal spray treatment or were observed only without nasal spray treatment. Participants who opted OL treatment phase received esketamine 56 mg nasal spray on Day 28 regardless of the treatment assignment in the DB phase and received subsequent doses at the same or adjusted (56 mg or 84 mg) dose level based on efficacy and tolerability with dosing frequency: twice weekly from Weeks 5 to 8 followed by once weekly from Weeks 9 to 12 and then weekly or every other week from Weeks 13 to 16 based on clinical judgment and was individualized to the least frequent dosing to maintain remission/response. During this period participants were given the option to receive standard-of-care treatment for depression. As planned, OL phase adverse events analysis was performed by treatment groups assigned in the DB phase, irrespective of the OL phase adjusted doses.
- OL Observation Period: After completion of DB treatment phase, participants who opted OL observation phase were only observed without esketamine nasal spray treatment but received standard-of-care treatment for depression.
- Follow up: All Participants: Participants who received at least 1 dose of study treatment in the DB or OL treatment phase entered into 1- week follow-up phase after their last dose of study treatment.
Arm/Group | DB: Placebo | DB: Esketamine 56 mg | DB: Esketamine 84 mg | OL Treatment: Placebo to Esketamine | OL Treatment: Esketamine 56 mg to Esketamine | OL Treatment: Esketamine 84 mg to Esketamine | OL Observation Period | Follow up: All Participants
All-Cause Mortality (participants affected / at risk) | 0/250 | 0/106 | 0/121 | 0/237 | 0/99 | 0/105 | 0/1 | 0/477
Serious Adverse Events (participants affected / at risk) | 3/250 | 1/105 | 2/121 | 6/237 | 3/99 | 0/105 | 0/1 | 1/476
Other Adverse Events (participants affected / at risk) | 73/250 | 69/105 | 80/121 | 147/237 | 49/99 | 44/105 | 0/1 | 8/476
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Placebo (N=250) | DB: Esketamine 56 mg (N=105) | DB: Esketamine 84 mg (N=121) | OL Treatment: Placebo to Esketamine (N=237) | OL Treatment: Esketamine 56 mg to Esketamine (N=99) | OL Treatment: Esketamine 84 mg to Esketamine (N=105) | OL Observation Period (N=1) | Follow up: All Participants (N=476)
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Hernia Obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ophthalmic Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Self-Injurious Ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Placebo (N=250) | DB: Esketamine 56 mg (N=105) | DB: Esketamine 84 mg (N=121) | OL Treatment: Placebo to Esketamine (N=237) | OL Treatment: Esketamine 56 mg to Esketamine (N=99) | OL Treatment: Esketamine 84 mg to Esketamine (N=105) | OL Observation Period (N=1) | Follow up: All Participants (N=476)
Diarrhoea (Gastrointestinal disorders) | 6 | 3 | 1 | 16 | 5 | 3 | 0 | 1
Nausea (Gastrointestinal disorders) | 21 | 24 | 32 | 69 | 18 | 15 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 5 | 10 | 27 | 6 | 2 | 0 | 1
Fatigue (General disorders) | 11 | 8 | 7 | 18 | 6 | 5 | 0 | 0
Feeling Drunk (General disorders) | 2 | 8 | 8 | 13 | 6 | 6 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 2 | 12 | 0 | 1 | 0 | 4
Dizziness (Nervous system disorders) | 18 | 22 | 27 | 45 | 8 | 10 | 0 | 1
Dysgeusia (Nervous system disorders) | 9 | 5 | 5 | 14 | 4 | 5 | 0 | 0
Headache (Nervous system disorders) | 22 | 19 | 24 | 36 | 13 | 11 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 2 | 5 | 15 | 2 | 4 | 0 | 0
Somnolence (Nervous system disorders) | 4 | 6 | 3 | 10 | 2 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 5 | 10 | 14 | 3 | 4 | 0 | 0
Dissociation (Psychiatric disorders) | 7 | 23 | 32 | 42 | 12 | 15 | 0 | 0
Insomnia (Psychiatric disorders) | 9 | 6 | 5 | 9 | 2 | 1 | 0 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 4 | 13 | 2 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT04599855/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT04599855/SAP_001.pdf